CLINICAL TRIAL: NCT04480346
Title: Multisite Study of School-based Treatment Approaches for Adolescents With ADHD
Brief Title: Multisite Study of High School-based Treatment for Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: Lehigh University (Other)
Responsible Party: Principal Investigator, Steven Evans, Distinguished Professor of Psychology, Ohio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R305A140356 - 15
Record Dates: First submitted 2020-07-10; First posted 2020-07-21 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHP treatment (Experimental): Participants assigned to this arm received the treatment described in another section.
  Interventions: Behavioral: Challenging Horizons Program
- Community Care (No Intervention): Participants randomly assigned to this condition received information about service providers in the community, but no services from the investigators.

INTERVENTIONS:
Behavioral: Challenging Horizons Program — Intervention delivered in high schools provided by school mental health professional over the course of an academic year with twice-weekly meetings with students and 10 evening group meetings with students and 10 group sessions with parents.
  Arms: CHP treatment

SUMMARY:
We evaluated the extent to which receiving the school-based multi-component treatment of the Challenging Horizons Program (CHP) would lead to significant improvements in levels of symptoms of attention deficit hyperactivity disorder (ADHD) and social and academic functioning for high school aged adolescents diagnosed with ADHD. We intended to recruit 200 high school aged adolescents with a diagnosis of ADHD who would be randomly assigned to either CHP or a Community Care condition within each of 12 participating high schools. Outcome measures included parent, teacher and adolescent reports as well as observational data. Measures were collected at initial evaluations which preceded the one academic year of treatment, during the treatment period, and at six-months after treatment ended. Based on previous research with this treatment in middle and high schools, we anticipated meaningful gains for those in the treatment condition at post-treatment and larger gains on some variables at the 6-month follow-up evaluation.

DETAILED DESCRIPTION:
We evaluated the extent to which receiving the school-based multi-component treatment of the Challenging Horizons Program (CHP) would lead to significant improvements in levels of symptoms of attention deficit hyperactivity disorder (ADHD) and social and academic functioning for high school aged adolescents diagnosed with ADHD. We intended to recruit 200 high school aged adolescents with a diagnosis of ADHD who would be randomly assigned to either CHP or a Community Care condition within each of 12 participating high schools. Outcome measures included parent, teacher and adolescent reports as well as observational data. Measures were collected at initial evaluations which preceded the one academic year of treatment, during the treatment period, and at six-months after treatment ended. Based on previous research with this treatment in middle and high schools, we anticipated meaningful gains for those in the treatment condition at post-treatment and larger gains on some variables at the 6-month follow-up evaluation. Eligible participants were stratified for medication status and sex following the completion of all eligibility assessments for each of 3 cohorts and were randomly assigned (within schools) to either the CHP or CC condition. Siblings were assigned together such that they would be in the same condition. All measures (except the achievement test which was given at eligibility and post-treatment assessment points) were administered on at least three occasions including pre-treatment (i.e., eligibility or baseline), post-treatment, and 6-month follow-up. Rating scales were completed online using REDCap (Harris et al., 2009) with the exception of the School Functioning Scale.

Participants randomized to the treatment group met with their coaches individually for approximately 15-20 minutes twice per week throughout the academic year, typically during lunch, study hall, or an elective class. Individual sessions included study skills, organization, problem solving, and interpersonal skills training. Ten, 90-minute group sessions were offered to adolescents and parents in the evenings and ran concurrently. The organization intervention occurred during each individual session. During initial sessions, students and coaches worked collaboratively to develop a system of organizing the student's binders or folders and tracking assignments in a daily planner or electronic calendar. Subsequent sessions included a binder and daily planner check in which the student's adherence to the system was recorded and then the student practiced addressing disorganization (e.g., put assignments in the correct folders, update planner). After meeting objective criteria for organization (e.g., at least 80% planner completion for two consecutive weeks), adolescents independently completed organization and planner checks under supervision by coaches.

Each month, coaches checked with students and school records regarding six areas of risk including tardiness, absenteeism, in-school disciplinary actions, out-of-school suspension, failing classes, and missing assignments. If students met a predetermined threshold for risk (e.g., 80% or fewer assignments turned in on time), then the student and coach had a problem-solving discussion. The goal was to both develop a solution to the relevant problem as well as teach students how to use problem-solving skills. The process included (1) defining the problem, (2) setting a goal, (3) brainstorming ways to achieve that goal, (4) selecting one or more of these solutions, (5) determining how to know if the plan is working, (6) setting a date to start implementation, and (7) setting a date to review the success of the plan. During a subsequent session, the coach and student reviewed the results of the plan relative to stated goals and determined if they should continue the plan or make changes. During individual sessions, students and coaches critically reviewed social events and the student's behavior in relation to goals. This was an extension of the evening sessions focused on ISG and involved applying the skills learned in the group meetings to individual social events in the participants' daily lives. For students who were not performing well on tests and quizzes, coaches provided study skills intervention. Coaches reviewed test-taking strategies regarding different styles of test questions (e.g., planning an outline for an essay question). Students were tested on these strategies to demonstrate mastery and then practice the skills on practice tests. Students also learned strategies for using flashcards and class notes effectively to prepare for tests. In the ten evening sessions offered for students the adolescents participated in an interpersonal skills group (ISG) to improve social skills. During the first group, students were introduced to the concepts of ideal self - how they want to be seen, and real self - how they really are seen. Students developed ideal self goals and practiced behaving in ways that aligned with these goals during games and activities and frequently reviewed progess with staff. Parents were offered 10 evening sessions concurrent with students' ISG. Program staff provided psychoeducation about ADHD and common difficulties faced by teenagers, including sleep hygiene. Parents also worked with project staff to develop a homework management plan that determined when students would complete homework each night and for how long.

Participants who were randomized to the CC condition were given a list of available resources in their community and received no services from research staff. Participants in both CC and the treatment condition were informed that they could receive any community services during the duration of the trial.

ELIGIBILITY:
Inclusion Criteria:

* On phone screen with parent report a previous diagnosis of ADHD or elevated levels on at least 4 of 9 ADHD symptoms of inattention
* Meet diagnostic criteria for ADHD on structured diagnostic interview with parents or parent and teacher ratings of symptoms and impairment
* Demonstrate an IQ of 75 or greater on the Wechsler Abbreviated Scale of Intelligence - Second Edition
* Attend a participating high school

Exclusion Criteria:

* Does not exceed critical threshold on adolescent self report of substance us on the Substance Abuse Subtle Screening Inventory
* Does not meet diagnostic criteria for bipolar disorder, psychosis, or obsessive-compulsive disorder

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
ADHD symptoms | Change from Baseline ADHD symptoms through study completion, an average of 9 months.
  Parent ratings of 18 DSM symptoms of ADHD;The scores range from 0 to 54 with high scores representing worse symptoms.
ADHD symptoms | Change from Baseline ADHD symptoms through six months post treatment, an average of 15 months.
  Parent ratings of 18 DSM symptoms of ADHD;The scores range from 0 to 54 with high scores representing worse symptoms.
Social Skills | Change from Baseline social skills through study completion, an average of 9 months.
  Parent ratings on Social Skills Improvement System Rating Scale - parent rating version;There are 46 items on the social skills factor that are rated from 0 to 3 (range 0 to 138) with higher scores indicating better social skills. Scores are converted to age and sex based standard scores (M=100).
Social Skills | Change from Baseline social skills through six months post treatment, an average of 15 months.
  Parent ratings on Social Skills Improvement System Rating Scale - parent rating version;There are 46 items on the social skills factor that are rated from 0 to 3 (range 0 to 138) with higher scores indicating better social skills. Scores are converted to age and sex based standard scores (M=100).
Grade Point Average | Change from Baseline grade point average through study completion, an average of 9 months
  Average of grades assigned by school each grading period;Average calculated based on a 0 to 4 scale with higher GPA corresponding to higher grades.
Grade Point Average | Change from Baseline grade point average through six months post treatment, an average of 15 months.
  Average of grades assigned by school each grading period;Average calculated based on a 0 to 4 scale with higher GPA corresponding to higher grades.
Organization Skills | Change from Baseline organization skills through study completion, an average of 9 months.
  Parent ratings on the Children's Organization Skills Scale;This is a 66-item rating scale with three subscales including Task Planning (raw scores range from 6 to 24), Organizing Actions (raw scores range from 10 to 40), and Memory and Materials Management (raw scores range from 10 to 40). High scores indicate worse organization skills.
Organization Skills | Change from Baseline organization skills through six months post treatment, an average of 15 months.
  Parent ratings on the Children's Organization Skills Scale;This is a 66-item rating scale with three subscales including Task Planning (raw scores range from 6 to 24), Organizing Actions (raw scores range from 10 to 40), and Memory and Materials Management (raw scores range from 10 to 40). High scores indicate worse organization skills.
Homework Completion | Change from Baseline Homework Completion through study completion, an average of 9 months.
  Parent ratings on the Homework Problems Checklist;This is a 20 item scale with scores ranging from 0 to 60 and high scores indicate greater problems completing homework.
Homework Completion | Change from Baseline Homework Completion through six months post treatment, an average of 15 months.
  Parent ratings on the Homework Problems Checklist;This is a 20 item scale with scores ranging from 0 to 60 and high scores indicate greater problems completing homework.
Classroom Behavior and Academic Performance | Change from Baseline classroom behavior and academic performance through study completion, an average of 9 months.
  Teacher ratings on the School Functioning Scale;This is a 9-item scale designed to measure behavior and academic performance in secondary school classrooms with scores ranging from 9 to 47. One 4-item factor focuses on classroom engagement behaviors and performance on tests and quizzes and scores range from 4 to 20 with high scores indicating better performance. Three questions about disruptive behavior have a range of scores from 3 to 15 with high scores indicating more disruption. Two questions focusing on interpersonal relationships produce scores ranging from 2 to 12 with high scores indicating better relationships.
Classroom Behavior and Academic Performance | Change from Baseline classroom behavior and academic performance through six months post treatment, an average of 15 months.
  Teacher ratings on the School Functioning Scale;This is a 9-item scale designed to measure behavior and academic performance in secondary school classrooms with scores ranging from 9 to 47. One 4-item factor focuses on classroom engagement behaviors and performance on tests and quizzes and scores range from 4 to 20 with high scores indicating better performance. Three questions about disruptive behavior have a range of scores from 3 to 15 with high scores indicating more disruption. Two questions focusing on interpersonal relationships produce scores ranging from 2 to 12 with high scores indicating better relationships.

SECONDARY OUTCOMES:
Emotion Regulation | Change from Baseline emotion regulation through study completion, an average of 9 months.
  Student ratings on the Difficulties with Emotion Regulation Scale;This is a 36-item scale with scores ranging from 0 to 180 and high scores representing more dysregulation of emotion.
Emotion Regulation | Change from Baseline emotion regulation through six months post treatment, an average of 15 months.
  Student ratings on the Difficulties with Emotion Regulation Scale;This is a 36-item scale with scores ranging from 0 to 180 and high scores representing more dysregulation of emotion.
Anxiety | Change from Baseline anxiety through study completion, an average of 9 months.
  Student ratings on the Beck Youth Inventory II;This is a 20-item scale ranging from 0 to 80 with high scores representing more anxiety.
Anxiety | Change from Baseline anxiety through six months post treatment, an average of 15 months.
  Student ratings on the Beck Youth Inventory II;This is a 20-item scale ranging from 0 to 80 with high scores representing more anxiety.
Depression | Change from Baseline depression through study completion, an average of 9 months.
  Student ratings on the Reynold's Adolescent Depression Scale 2 - Short Form:This is a 10-item measure with item scores ranging from 1 to 4 (total range 10 to 40) and higher scores indicate greater depression.
Depression | Change from Baseline depression through six months post treatment, an average of 15 months.
  Student ratings on the Reynold's Adolescent Depression Scale 2 - Short Form;This is a 10-item measure with item scores ranging from 1 to 4 (total range 10 to 40) and higher scores indicate greater depression.
School Performance | Change from Baseline school performance through study completion, an average of 9 months.
  Parent ratings on the Adolescent Academic Problems Checklist;This is a 24-item checklist with scores ranging from 0 to 72 and high scores indicating greater problems.
School Performance | Change from Baseline school performance through six months post treatment, an average of 15 months.
  Parent ratings on the Adolescent Academic Problems Checklist;This is a 24-item checklist with scores ranging from 0 to 72 and high scores indicating greater problems.
Symptoms of conduct disorder and oppositional defiant disorder | Change from Baseline symptoms of conduct disorder and oppositional defiant disorder through study completion, an average of 9 months.
  Parent ratings on the Disruptive Behavior Disorders checklist;This is a 23-item scale with scores ranging from 0 to 69 with high scores indicating a higher level of symptoms.
Symptoms of conduct disorder and oppositional defiant disorder | Change from Baseline symptoms of conduct disorder and oppositional defiant disorder through six months post treatment, an average of 15 months.
  Parent ratings on the Disruptive Behavior Disorders checklist;This is a 23-item scale with scores ranging from 0 to 69 with high scores indicating a higher level of symptoms.
Family relationships | Change from Baseline family relationships through study completion, an average of 9 months.
  Parent ratings on the Index of Family Relations;This is a 25-item scale with scores ranging from 0 to 150 with high scores indicating greater family distress in relationships.
Family relationships | Change from Baseline family relationships through six months post treatment, an average of 15 months.
  Parent ratings on the Index of Family Relations;This is a 25-item scale with scores ranging from 0 to 150 with high scores indicating greater family distress in relationships.
Parent stress | Change from Baseline parent stress through study completion, an average of 9 months
  Parent ratings on the Stress Index for Parents of Adolescents;This is a 112-item scale and we used the 40-item Adolescent Domain subscale and the 32-item Adolescent-Parent Relationship Domain scale. Scores on the Adolescent Domain subscale ranged from 40 to 200 and scores on the Adolescent-Parent Relationship Domain scale ranged from 32 to 160 with high scores on each scale reflecting greater parent stress.
Parent stress | Change from Baseline parent stress through six months post treatment, an average of 15 months.
  Parent ratings on the Stress Index for Parents of Adolescents;This is a 112-item scale and we used the 40-item Adolescent Domain subscale and the 32-item Adolescent-Parent Relationship Domain scale. Scores on the Adolescent Domain subscale ranged from 40 to 200 and scores on the Adolescent-Parent Relationship Domain scale ranged from 32 to 160 with high scores on each scale reflecting greater parent stress.
Academic Achievement | Change from Baseline academic achievement through study completion, an average of 9 months.
  Adolescent's performance on the Woodcock Johnson Tests of Achievement;This is a comprehensive performance measure of achievement with standard scores with a mean of 100 and higher scores indicating higher levels of achievement.
Academic Achievement | Change from Baseline academic achievement through six months post treatment, an average of 15 months.
  Adolescent's performance on the Woodcock Johnson Tests of Achievement;This is a comprehensive performance measure of achievement with standard scores with a mean of 100 and higher scores indicating higher levels of achievement.

CONTACTS AND LOCATIONS:
Overall Officials: Steven W Evans, Ph.D., Principal Investigator — Ohio University
Locations (2):
- United States (2):
  - Ohio University, Athens, Ohio
  - Lehigh University, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available after the main outcome studies are published. The Co-PIs will consider requests in relation to potential overlap with investigator team planned manuscripts and qualifications of person making the request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after main outcome studies are published.
Access Criteria: Contact either of the Co-PIs (Evans & DuPaul)

REFERENCES:
- [Background] Dawson AE, Wymbs BT, Evans SW, DuPaul GJ. Exploring how adolescents with ADHD use and interact with technology. J Adolesc. 2019 Feb;71:119-137. doi: 10.1016/j.adolescence.2019.01.004. Epub 2019 Jan 25. PMID 30690333
- [Background] DuPaul GJ, Evans SW, Allan D, Puzino K, Xiang J, Cooper J, Owens JS. High school teacher ratings of academic, social, and behavioral difficulties: Factor structure and normative data for the School Functioning Scale. Sch Psychol. 2019 Sep;34(5):479-491. doi: 10.1037/spq0000323. Epub 2019 May 2. PMID 31045408
- [Background] Bunford N, Dawson AE, Evans SW, Ray AR, Langberg JM, Owens JS, DuPaul GJ, Allan DM. The Difficulties in Emotion Regulation Scale-Parent Report: A Psychometric Investigation Examining Adolescents With and Without ADHD. Assessment. 2020 Jul;27(5):921-940. doi: 10.1177/1073191118792307. Epub 2018 Aug 16. PMID 30112924
- [Background] Margherio SM, Capps ER, Monopoli JW, Evans SW, Hernandez-Rodriguez M, Owens JS, DuPaul GJ. Romantic Relationships and Sexual Behavior Among Adolescents With ADHD. J Atten Disord. 2021 Aug;25(10):1466-1478. doi: 10.1177/1087054720914371. Epub 2020 Apr 24. PMID 32329399
- [Background] Margherio SM, Brickner MA, Evans SW, Sarno Owens J, DuPaul GJ, Allan NP. The role of emotion regulation in alcohol use among adolescents with attention-deficit/hyperactivity disorder. Psychol Addict Behav. 2020 Nov;34(7):772-782. doi: 10.1037/adb0000582. Epub 2020 Apr 9. PMID 32271054
- [Background] Monopoli WJ, Evans SW, Benson K, Allan NP, Owens JS, DuPaul GJ, Bunford N. Assessment of a conceptually informed measure of emotion dysregulation: Evidence of construct validity vis a vis impulsivity and internalizing symptoms in adolescents with ADHD. Int J Methods Psychiatr Res. 2020 Dec;29(4):1-14. doi: 10.1002/mpr.1826. Epub 2020 Sep 8. PMID 32898309
- [Background] Hustus, C., Evans, S.W., Owens, J.S., Benson, K.E., Hetrick, A., Kipperman, K. & DuPaul, G.J. (in press). An evaluation of 504 and individualized educational programs for high school students with attention-deficit/hyperactivity disorder. School Psychology Review.
- [Background] Cleminshaw CL, DuPaul GJ, Kipperman KL, Evans SW, Owens JS. Social deficits in high school students with attention-deficit/hyperactivity disorder and the role of emotion dysregulation. Sch Psychol. 2020 Jul;35(4):233-242. doi: 10.1037/spq0000392. PMID 32673052
- [Derived] DuPaul GJ, Evans SW, Cleminshaw-Mahan CL, Fu Q. School-Based Intervention for Adolescents With ADHD: Predictors of Effects on Academic, Behavioral, and Social Functioning. Behav Ther. 2024 Jul;55(4):680-697. doi: 10.1016/j.beth.2024.01.010. Epub 2024 Feb 13. PMID 38937043
- [Derived] Evans SW, DuPaul GJ, Benson K, Owens JS, Fu Q, Cleminshaw C, Kipperman K, Margherio S. Social Functioning Outcomes of a High School-Based Treatment Program for Adolescents with ADHD. J Clin Child Adolesc Psychol. 2024 May-Jun;53(3):413-428. doi: 10.1080/15374416.2023.2235693. Epub 2023 Jul 26. PMID 37494306